CLINICAL TRIAL: NCT03502421
Title: A Randomized Controlled Trial to Determine the Efficacy of Ketamine as an Adjunct for Pain Management in Patients With Sickle Cell Crisis
Brief Title: Ketamine Sickle Cell Disease
Acronym: SCD
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Never IRB approved, no intention to proceed with the study
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00033576
Record Dates: First submitted 2018-04-10; First posted 2018-04-18 (Actual); Last update posted 2018-09-26 (Actual); Status verified 2018-04

CONDITIONS: SC Disease; Pain, Chronic
Keywords: Ketamine
MeSH Terms: conditions — Hemoglobin SC Disease; Chronic Pain | interventions — Ketamine

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Prospective Clinical Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ketamine (Experimental): Continuous infusion of Ketamine 0.3 to 0.5 mg/kg per hour PCA Dilaudid 2.0-2.5 mg
  Interventions: Drug: Ketamine
- Opioid Only (No Intervention): Patient-controlled analgesia Dilaudid 2.0-2.5 mg

INTERVENTIONS:
Drug: Ketamine — Low dose continuous infusion of ketamine 0.3 to 0.5 mg/kg per hour
  Arms: Ketamine

SUMMARY:
Sickle cell disease (SCD) often results in acute vaso-occlusive crisis (VOC), an obstruction of blood vessels resulting in ischemic injury and pain. The pain experienced during these episodes is due to a wide range of pathophysiological processes. Though recent studies have begun to unravel the underlying mechanisms of these processes, literature focused on pain management for sickle cell disease is scarce. Opioids and non-steroidal anti-inflammatory drugs (NSAIDs) remain the predominate treatment for VOC.

However, the efficacy of these treatments has come into question. A large sub-set of patients with SCD report continued pain despite treatment with opioids. Tolerance and opioid-induced hyperalgesia (OIH) may be responsible for unresponsiveness to opioid-centric treatment modalities. New classes of drugs are being tested to prevent and treat acute pain associated with SCD, but in the meantime physicians are looking to existing therapies to bridge the gap.

The N-methyl-d-aspartate (NMDA) receptor has been implicated in both tolerance and OIH. As a NMDA receptor agonist, ketamine has been shown to modulate opioid tolerance and OIH in animal models and clinical settings. Ketamine utilized as a low dose continuous infusion could benefit patients with SCD related pain that are unresponsive to opioid analgesics. Based on limited studies of adjuvant ketamine use for pain management, low-dose ketamine continuous infusion appears safe. Further clinical investigations are warranted to fully support the use of low-dose ketamine infusion in patients with SCD-related pain.

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed with sickle cell anemia
* Adults aged 18 and older
* Subjects who have given written consent

Exclusion Criteria:

* Subjects who are pregnant
* Subjects younger than 18 years
* Subjects known or suspected to have an allergy to opiates/opioids, muscle relaxants or other similar medications
* Subjects who have a contraindication to ketamine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2019-09-01 (Estimated); Study Completion 2019-11-01 (Estimated)

PRIMARY OUTCOMES:
Total opioid Use in milligrams morphine equivalents | 1-3 hours
  Total opioid Use in milligrams morphine equivalents
Pain scores measured on the Visual Analog Scale 0 - 10 | 1-3 hours
  Pain scores measured on the Visual Analog Scale 0 - 10

SECONDARY OUTCOMES:
Cost of pharmacotherapy | 1 day
  monetary cost of intervention used
Length of hospital stay | 1-7 days
  Length of stay in the hospital
Nausea and vomiting scores Visual Analog Scale 0 - 10 | 1-3 hours
  Nausea and vomiting scores Visual Analog Scale 0 - 10

CONTACTS AND LOCATIONS:
Overall Officials: Enrico Camporesi, MD, Principal Investigator — University of South Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Puri L, Nottage KA, Hankins JS, Anghelescu DL. State of the Art Management of Acute Vaso-occlusive Pain in Sickle Cell Disease. Paediatr Drugs. 2018 Feb;20(1):29-42. doi: 10.1007/s40272-017-0263-z. PMID 28853040
- [Background] Neri CM, Pestieau SR, Darbari DS. Low-dose ketamine as a potential adjuvant therapy for painful vaso-occlusive crises in sickle cell disease. Paediatr Anaesth. 2013 Aug;23(8):684-9. doi: 10.1111/pan.12172. Epub 2013 Apr 9. PMID 23565738
- [Background] Visser E, Schug SA. The role of ketamine in pain management. Biomed Pharmacother. 2006 Aug;60(7):341-8. doi: 10.1016/j.biopha.2006.06.021. Epub 2006 Jul 5. PMID 16854557
- [Background] Aguado D, Abreu M, Benito J, Garcia-Fernandez J, Gomez de Segura IA. Ketamine and remifentanil interactions on the sevoflurane minimum alveolar concentration and acute opioid tolerance in the rat. Anesth Analg. 2011 Sep;113(3):505-12. doi: 10.1213/ANE.0b013e318227517a. Epub 2011 Jul 21. PMID 21778336
- [Background] Sun J, Lin H, Feng X, Dong J, Ansong E, Xu X. A comparison of intrathecal magnesium and ketamine in attenuating remifentanil-induced hyperalgesia in rats. BMC Anesthesiol. 2016 Sep 6;16(1):74. doi: 10.1186/s12871-016-0235-9. PMID 27599837